CLINICAL TRIAL: NCT00217100
Title: Folic Acid for Vascular Outcome Reduction in Transplantation.
Brief Title: A Multivitamin Comparison Study in Kidney Transplant Recipients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Wisconsin, Madison (Other); University of California, San Francisco (Other); University of Alabama at Birmingham (Other); Ohio State University (Other)
Responsible Party: Fernando G Cosio, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1965-04
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Kidney Transplant Recipients
MeSH Terms: interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Multi Vitamin Formulation (Active Comparator)
  Interventions: Dietary Supplement: Multivitamin
- Sugar pill (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Multivitamin — 1 tablet a day
  Arms: Multi Vitamin Formulation
Dietary Supplement: Placebo — 1 tablet a day
  Arms: Sugar pill

SUMMARY:
This study is being done to compare arteriosclerotic cardiovascular disease in kidney transplant recipient taking a standard multivitamin versus those taking a multivitamin augmented by a high dose combination of folic acid, vitamin B12, and vitamin B6.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind controlled clinical trial. The trial has been designed to determine whether total homocysteine lowering treatment with a standard multivitamin augmented by a multivitamin containing no folic acid B12, and vitamin B6, versus treatment with an identical multivitamin containing no folic acid, will reduce the pooled rate of recurrent or new cardiovascular disease outcomes or events. Participants will have a brief visit, at which the participant will have physical measurements, blood pressure and history taken. Urine and blood tests will be performed to determine the levels of homocysteine, vitamins and creatinine. Qualifying participants will be randomly assigned to receive multivitamins containing a high dose of folic acid, vitamin B6, and vitamin B12, or an identical multivitamin containing no folic acid, and estimated average requirement amounts of vitamin B6 and vitamin B12. The participant will be required to return annually throughout the next five years for physical exams, blood and urine tests.

ELIGIBILITY:
Participants with elevated homocysteine levels that are between the ages of 35-75 years old and have had a kidney transplant with stable renal graft function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Estimated Average Requirement (EAR) amounts | basline to death or common end date 4.5 years
  to determine whether total homocysteine (tHcy)-lowering treatment with a standard multivitamin augmented by a high dose combination of folic acid, vitamin B12, and vitamin B6, versus treatment with an identical multivitamin containing no folic acid, and Estimated Average Requirement (EAR) amounts of vitamin B6 and vitamin B12., reduces the pooled rate of recurrent and de novo cardiovascular disease [CVD]outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States